CLINICAL TRIAL: NCT04296708
Title: The Influence of a Ten-week ExerCube Training on Executive Functions as Well as on Training Motivation, Enjoyment and Mental Well-being in Young Athletes
Brief Title: ExerCube Training on Executive Functions in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EK 2019-N-161
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-03

CONDITIONS: Effects of Exergaming on Cognitive Functions in Young Athleten
Keywords: Exergaming; Cognitive Functions; Young athletes; Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ExerCube group (Experimental): The ExerCube is an immersive fitness game setting that combines innovative soft- and hardware designs with state of-the-art training concepts. The ExerCube has three walls which serve as virtual reality projection screens and haptic interfaces. The ExerCube is a playful physical-cognitive exergame training. The user navigates a virtual environment/reality via whole body exercise. The video game navigates the user and triggers various cognitive functions. The used physical exercises are functionally and elicit the improvement of endurance and strength components. Via different monitoring systems (points and heart rate), the game adapts to the individual abilities and training level to tailor workout intensity. The ExerCube training consists of two sessions a week each session will last about 30 minutes of which 25 minutes will be pure playtime
  Interventions: Other: Exergame Training
- Control group (No Intervention): The control group does not have any additional ExerCube training.

INTERVENTIONS:
Other: Exergame Training — An exergame combines exercise and gaming in a holistic approach.
  Arms: ExerCube group

SUMMARY:
Competitive game sports require the existence of several sport-specific skills. In particular, game sport athletes need a good set of skills in order to perform well on the field. Therefore, it is important for athletes, especially young athletes, not only perform their sport, but also perform variable trainings, which differently train/trigger sport-specific skills. One skill set that is important in competitive game sports are so-called executive functions. Executive functions are needed for action planning and adaptation to the individual environmental situation, e.g. inhibition, flexibility and divided attention. A form of training that is very promising in this respect is exergaming as nowadays coaches are using virtual reality simulations to create realistic training environments. An exergame that combines this cognitive stimulation with whole-body movements in a motivating training environment is the ExerCube. Until now, however, evidence is lacking how an additional holistic exergame training can influence executive functioning in young athletes. Therefore, this study aims to get preliminary insight into the effects of the ExerCube performance on the executive function in young athletes (primary objective). The participants will be allocated into either the intervention group (ExerCube training) or the control group (no additional ExerCube training). The intervention group will train 2 times per week for about 30 minutes over a time frame of 10 weeks. Additionally, to consider the effects of the training environment, the secondary objectives include training motivation, enjoyment and flow as well as mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* Age between 15 to 20 years
* Young athletes (game sports)
* Healthy (self-reported)
* Able to provide written informed consent and understand instructions

Exclusion Criteria:

* History of cardiovascular issue that would prevent training participation
* Asthma (not controllable)
* Musculosceletal injuries that would prevent training participation
* Pain that would be reinforced by sportive activities
* Pregnancy

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
FitLight | Before and after the intervention, within two weeks
  FitLight Trainer™ (Sports Corp. Ontario, Canada) is a commercially available product and consists of eight LED powered lights controlled by a wireless connection via a tablet. The tablet is running on android version 4.2.2 and has in advance a FitLight Trainer™ software to interact with the lights. With this software, it is possible to generate new specific light sequences.The FitLight allow the testing of executive functions depending on the programmed sequences. The participants use whole-body movements of arms and legs to solve the programmes sequences. Before the participants execute the main test, they perform a pre-test to minimize the learning effect and to get familiar with the test environment
Test for Attentional Performance | Before and after the intervention, within two weeks
  Initially the TAP (D-TAP 2.3 VL, PSYTEST, Psychologische Testsysteme, Herzogenrath, Germany) was developed to assess attentional deficits in a cerebral impaired population. The participants perform a simple reaction task.The stimuli are presented on a screen of a personal computer. Before the participants execute the main test, they perform a pre-test to minimize the learning effect and to get familiar with the test environment.

SECONDARY OUTCOMES:
Situation Motivation Scale | Before and after the intervention, within two weeks
  The Situation Motivation Scale was designed to assess the constructs of intrinsic motivation, identified regulation, external regulation and amotivation in field and laboratory settings.
  - 16 items graded on a 7-point Likert scale, a higher score means a better outcome
Flow Short Scale | Before and after the intervention, within two weeks
  The first 10 items measure the components of Flow-Experience as first described by Mihaly Csikszentmihalyi 1975. The items 11 - 13 measure Worry someone may have in the situation the measurement is made.
  - 13 items graded on a 7-point Likert scale, Item 1-10: a higher score means a better outcome, Item 11-13: a lower score means a better outcome
Physical Activity Enjoyment Scale | Before and after the intervention, within two weeks
  The Physical Activity Enjoyment Scale was developed to measure physical activity enjoyment using college-aged students. The scale is a reliable and valid measure of enjoyment in physical activity environments.
  - 18 bipolar statements and a 7-point continuum, a higher score means a better outcome
Warwick-Edinburgh Mental Well-being Scale | Before and after the intervention, within two weeks
  This mental well-being scale is a valid measurement at a population and on an individual level. The questionnaire consists of 14 items and covers following aspects of mental health: positive affect (feelings of optimism, cheerfulness, and relaxation), satisfying interpersonal relationships, positive functioning (energy, clear thinking, self-acceptance, personal development, competence and autonomy). A minimum score of 14 and a maximum score of 70 can be achieved, whereas a score from 51 can be assumed normal. The higher the score is, the higher the level of mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided